CLINICAL TRIAL: NCT00573261
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Center Study Designed to Assess the Effects of Pregabalin on Change in Patients With Diabetic Neuropathy
Brief Title: A Randomized Double-Blind Study Testing the Effects of Pregabalin on Diabetic Neuropathy
Acronym: Pregabalin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00009557; 2005-0003 (Other: Pfizer); 7511-05-8 (Other: Duke legacy protocol number)
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Results first posted 2013-07-18 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2013-07

CONDITIONS: Diabetic Neuropathy
Keywords: Diabetic neuropathy; Pregabalin; Lyrica
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregabalin (Experimental): Pregabalin medication
  Interventions: Drug: Pregabalin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — Subjects will take pregabalin for the duration of four weeks. The dosage will range from 75 mg twice a day to 300 mg twice a day.
  Other Names: Lyrica
  Arms: Pregabalin
Drug: Placebo — Subjects will take placebo for the duration of four weeks. The dosage will range from 75 mg twice a day to 300 mg twice a day.
  Arms: Placebo

SUMMARY:
This study is designed to examine how pregabalin affects parameters of autonomic nerve regulation in correlation with change in pain, anxiety, and depressive symptoms in patients with diabetic neuropathy.

DETAILED DESCRIPTION:
This study is designed to primarily examine how pregabalin affects the autonomic nerve or sympathetic-parasympathetic regulation in patients with diabetic neuropathy and its relationship to neuropathic pain. The goals of this study include (1) assessing the change of parameters of autonomic nerve function such as heart rate variability (HRV), respiratory sinus arrhythmia (RSA), minute ventilation, and changes in objective sleep parameters measured by means of the LifeShirt, upon treatment of pregabalin in comparison to placebo; (2) assessing the symptom change of neuropathic pain upon treatment of pregabalin in comparison to placebo; (3) assessing the change of anxiety symptoms upon treatment of pregabalin in comparison to placebo; (4) assessing the change of depressive symptoms upon treatment of pregabalin in comparison to placebo; (5) assessing the relationship of autonomic nerve function with neuropathic pain at baseline prior to treatment and the correspondences to the study drug; (6) assessing the relationship of autonomic nerve function with anxiety and depressive symptoms at baseline prior to treatment and their correspondences to the study drug; (7) identifying sensitive and reliable parameters of autonomic nerve regulation as predictor(s) of the severity and improvement of neuropathic pain and/or anxiety; and (8) to assess the change in objective sleep parameters (EEG/EOG) by means of the LifeShirt, upon treatment of pregabalin in comparison to placebo

ELIGIBILITY:
Inclusion Criteria:

* Outpatients aged 18 years or older
* Meet criteria for diagnosis of diabetic neuropathy
* Average daily pain scores greater than or equal to 4 by Visual Analog Scale
* Ability to give informed consent
* No pregnancy

Exclusion Criteria:

* Patients with clinically significant psychiatric disorders requiring vigorous interventions, i.e., moderate to severe depressive disorder, psychotic disorders, PTSD, obsessive compulsive disorder, panic disorder, substance abuse, or personality disorders, or active suicidal/homicidal ideations, or past history of active suicidal ideation and/or attempts
* Patients on gabapentin which cannot be discontinued, meaning a dose greater than 1200mg. If a patient is on a dose of gabapentin that is less than 1200mg and he or she is willing to stop taking the medication, he or she can participate in the study. These patients must take the last dose of gabapentin the night before starting the study.
* Patients being non-compliant with diabetic control
* Inability to wear the LifeShirt
* Unable to participate or answer questions using a personal digital assistant input device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Jiang, M.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Jiang W, Ladd S, Martsberger C, Feinglos M, Spratt SE, Kuchibhatla M, Green J, Krishnan R. Effects of pregabalin on heart rate variability in patients with painful diabetic neuropathy. J Clin Psychopharmacol. 2011 Apr;31(2):207-13. doi: 10.1097/JCP.0b013e31820f4f57. PMID 21346609

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the outpatient endocrine clinics of a tertiary academic center and locally via advertisement between March 3, 2006 and April 1, 2008.
Pre-assignment Details: There were 4 subjects who provided study consent but did not complete the baseline assessment because of unwillingness to wear the LifeShirt monitor (n=2 in placebo arm) and inability of keeping baseline assessment appointment due to job reassignment (n=2 in pregabalin arm).
Groups:
- Placebo: Placebo
  Placebo : Subjects will take placebo for the duration of four weeks. The dosage will range from 75 mg twice a day to 300 mg twice a day.
- Pregabalin: Pregabalin medication
  Pregabalin : Subjects will take pregabalin for the duration of four weeks. The dosage will range from 75 mg twice a day to 300 mg twice a day.
Period: Overall Study
Arm/Group | Placebo | Pregabalin
Started | 20 | 20
Completed | 14 | 15
Not Completed | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 13 | 29
  >=65 years | 4 | 7 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (14.36) | 59.65 (12.5) | 57.4 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 11 | 14 | 25
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Assessing the Change in Resting Blood Pressure Upon Treatment of Pregabalin vs. Placebo in Patients With Diabetes and Peripheral Neuropathy.
Time Frame: baseline and at end of a 4-week intervention
Population: A data card failure of the baseline heart rate record with the VivoMetrics system occurred for one subject who had completed baseline and 4-week assessments, leaving 28 subjects (n=13 in placebo, n=15 in pregabalin)having both completed baseline and end of 4-week R-R intervals for heart rate variability analysis.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Pregabalin: Pregabalin
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 13 | 15
mm Hg
  Systolic Blood Pressure (mm Hg) | -7.63 (10.46) | -8.98 (17.61)
  Diastolic Blood Pressure (mm Hg) | -4.41 (7.79) | -4.93 (8.64)

2. Secondary Outcome: To Assess the Change of Pain Symptoms Upon Treatment of Pregabalin in Comparison to Placebo.
Description: Pain severity was evaluated using the Visual Analog Scale, the Modified Brief Pain Inventory-Short Form, and the Neuropathy Pain Scale. The Visual Analog Scale was scored within a range of 0-100 with 0=no pain and 100=the worst imaginable pain. The Brief Pain Inventory is made up of two parts: total pain and pain interference. The total pain score is the sum of most, least, average, and now pain scored within a range of 0-10 with 0=no pain and 10=pain as bad as you can imagine. The pain interference score is the sum of affective and activity interference - how pain interfered with general activity, mood, walking ability, normal work, relationships, sleep, and enjoyment of life. It was scored within a range of 0-10 with 0=pain does not interfere and 10=pain completely interferes. The Neuropathy Pain Scale total is the sum of 10 items -cold, sharp, deep, dull, hot, intense, itchy, sensitive, surface, and unpleasant pain scored within a range of 0-10 with 0=no pain and 10=most pain.
Time Frame: baseline and end of 4 week intervention
Population: A data card failure of the baseline heart rate record with the VivoMetrics system occurred for one subject who had completed baseline and their 4-week assessments, leaving 28 subjects (n=13 in placebo, n=15 in pregabalin)having both completed baseline and end of 4-week R-R intervals for heart rate variability analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 13 | 15
units on a scale
  Visual analog pain rating | -21.29 (35.62) | -43.27 (32.03)
  Brief pain inventory - Total Pain | -1.36 (9.01) | -9.13 (9.63)
  Brief pain inventory - Most Pain | -1.07 (3.69) | -3.33 (3.46)
  Brief pain inventory - Least Pain | -0.071 (1.54) | -1.20 (1.93)
  Brief pain inventory - Average Pain | -0.64 (2.79) | -2.87 (3.04)
  Brief pain inventory - Now pain | 0.43 (1.95) | -1.73 (2.55)
  Pain interference | -1.43 (7.54) | -13.93 (10.35)
  Affective interference | -0.071 (3.69) | -5.27 (5.71)
  Activity Interference | -1.36 (4.94) | -8.67 (7.03)
  Neuropathy pain scale (total) | -10.31 (11.15) | -27.33 (22.95)
  Cold pain | -1.23 (3.37) | -2.13 (3.85)
  Sharp pain | -0.92 (2.40) | -2.53 (4.16)
  Deep pain | -0.23 (3.54) | -3.00 (3.51)
  Dull pain | 0 (2.38) | -2.07 (3.75)
  Hot pain | -1.77 (4.07) | -2.53 (3.40)
  Intense pain | -1.38 (1.66) | -3.13 (3.09)
  Itchy pain | 0 (2.08) | -4.07 (3.92)
  Sensitive pain | -2.31 (3.07) | -1.60 (3.11)
  Surface pain | -1.46 (1.56) | -3.20 (3.19)
  Unpleasant pain | -1.00 (2.38) | -3.07 (3.52)

3. Primary Outcome: Assessing the Change in Heart Rate by Means of the LifeShirt System Upon Treatment of Pregabalin vs. Placebo in Patients With Diabetes and Peripheral Neuropathy.
Description: The LifeShirt System, developed by VivoMetrics, is a lightweight vest with embedded sensors that continuously collect information on a range of cardiopulmonary parameters. It was used to collect and store the respiratory rate, posture, activity level, QRS complexes, and R-R intervals via a 3-axis accelerometer and a 3-lead, single channel electrocardiogram.
Time Frame: baseline and at end of a 4-week intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Beats Per Minute
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 13 | 15
Beats Per Minute | -2.94 (6.96) | -3.49 (5.51)

4. Primary Outcome: Assessing the Change in Heart Rate Variability by Means of the LifeShirt System Upon Treatment of Pregabalin vs. Placebo in Patients With Diabetes and Peripheral Neuropathy.
Description: Heart rate variability parameters generated by the frequency domain analysis included: total power (area under the curve) over all frequencies, very low frequency (VLF, 0-0.04 Hz),low frequency (LF, 0.04-0.15 Hz), and high frequency (HF,0.15-0.4 Hz).
Time Frame: baseline and at end of a 4-week intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hertz (Hz)
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 13 | 15
Hertz (Hz)
  Total Power | 45.29 (418.09) | -140.99 (629.81)
  Low Frequency | 32.41 (229.51) | -67.06 (252.06)
  High Frequency | -12.19 (79.91) | -41.37 (175.89)

5. Primary Outcome: Assessing the Change in Heart Rate Variability by Means of the LifeShirt System Upon Treatment of Pregabalin vs. Placebo in Patients With Diabetes and Peripheral Neuropathy.
Description: Heart Rate Variability parameters generated by the frequency domain analysis included: Low Frequency / High Frequency (LF/HF), as well as normalized LF (normalized LF=LF/[total power-VLF]) and normalized HF (normalized HF=HF/[total power-VLF]).
Time Frame: baseline and at end of a 4-week intervention
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- Pregabalin: Pregabalin
  Pregabalin : Subjects will take pregabalin for the duration of four weeks. The dosage will range from 75 mg twice a day to 300 mg twice a day.
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 13 | 15
Ratio
  Low frequency/High frequency | 0.37 (0.33) | -1.30 (2.89)
  Normalized low frequency | 0.0066 (0.023) | -0.049 (0.092)
  Normalized high frequency | -0.038 (0.066) | 0.039 (0.094)

6. Primary Outcome: Assessing the Change of Parameters of Autonomic Nerve Function Such as Heart Rate Variability by Means of the LifeShirt System Upon Treatment of Pregabalin vs. Placebo in Patients With Diabetes and Peripheral Neuropathy.
Description: Heart rate variability parameters yielded by time domain analysis included the mean of all R-R intervals (ANN), standard deviation of all R-R intervals (SDNN), root mean square of successive differences (RMSSD), and standard deviation of the averages of R-R intervals for all 5-minute segments within the block (SDANN).
Time Frame: baseline and at end of a 4-week intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 13 | 15
milliseconds
  ANN | 21.47 (84.56) | 65.44 (108.95)
  SDNN | 3.42 (8.83) | -0.55 (20.03)
  SDANN | 0.68 (7.67) | 1.38 (12.16)
  RMSSD | 0.58 (12.94) | -0.51 (8.44)

7. Primary Outcome: Assessing the Change of Parameters of Autonomic Nerve Function Such as Heart Rate Variability by Means of the LifeShirt System Upon Treatment of Pregabalin vs. Placebo in Patients With Diabetes and Peripheral Neuropathy.
Description: Heart rate variability parameters yielded by time domain analysis included the number of N-N intervals that differ by more than 50 milliseconds from adjacent intervals divided by the total number of all N-N intervals (pNN50).
Time Frame: baseline and at end of a 4-week intervention
Measure: Mean (Standard Deviation); unit: Intervals more than 50 ms
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 13 | 15
Intervals more than 50 ms | 15.97 (92.66) | -2.25 (41.81)

8. Primary Outcome: Assessing the Change of Parameters of Autonomic Nerve Function Such as Heart Rate Variability by Means of the LifeShirt System Upon Treatment of Pregabalin vs. Placebo in Patients With Diabetes and Peripheral Neuropathy.
Description: as for outcome 7
Time Frame: baseline and at end of a 4-week intervention
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 13 | 15
Ratio | 0.011 (0.087) | 0.0015 (0.051)

9. Secondary Outcome: To Assess the Change of Anxiety Symptoms Upon Treatment of Pregabalin in Comparison to Placebo.
Description: Anxiety symptoms were measured using the Spielberger State-Trait Anxiety Inventory Scale (STAI) for symptoms of anxiety. State anxiety: score range, 20-80 (higher score=greater levels of state anxiety). Trait anxiety: score range, 20-80 (higher score=greater levels of trait anxiety).
Time Frame: baseline and at end of a 4-week intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 13 | 15
units on a scale
  State Anxiety | 0.57 (5.91) | 1.2 (3.28)
  Trait Anxiety | 1 (6.16) | -3.67 (5.51)

10. Secondary Outcome: To Assess the Change of Depressive Symptoms Upon Treatment of Pregabalin in Comparison to Placebo.
Description: The Beck Depression Inventory Scale measures symptoms of depression, score range, 0-63 (higher score=greater severity of depressive symptoms)
Time Frame: baseline and at end of a 4-week intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 13 | 15
units on a scale | 1.21 (4.25) | -1.20 (1.57)

11. Secondary Outcome: To Assess the Change in Disability Scale Upon Treatment of Pregabalin in Comparison to Placebo.
Description: The Sheehan Disability Scale was used to evaluate functional impairment in work/school, social and family life, score range, 0-10; the 3 items can be summed into a single dimensional measure of global functional impairment that ranges from 0(unimpaired) to 30 (highly impaired).
Time Frame: baseline and at end of a 4-week intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 13 | 15
units on a scale
  Disability scale - Global functioning score | -1.67 (4.64) | -7.73 (7.70)
  Disability scale - Work/school disability | -0.42 (1.93) | -2.93 (3.26)
  Disability scale - Social disability | -0.58 (1.73) | -2.13 (2.83)
  Disability scale - Family disability | -0.67 (1.92) | -2.67 (3.02)

ADVERSE EVENTS:
Time Frame: Participants were contacted by phone starting at the end of week 1 for potential adverse effects and titration of the study drug throughout 4-week treatment period.
Arm/Group | Placebo | Pregabalin
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 0/14 | 3/15
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=14) | Pregabalin (N=15)
Dizziness (General disorders) | 0 (0) | 2 (2)
Swelling of the lower extremities (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study has a high dropout, which might have reduced the power of the analysis. One of the major reasons that many patients were not able to participate was an inability to commit to the relatively intense and frequent assessments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No